CLINICAL TRIAL: NCT02619162
Title: Nintedanib Plus Letrozole in Postmenopausal Women With Breast Cancer: Clinical Trial Phase 0/1 Safety and Pharmacodynamics
Brief Title: Nintedanib+Letrozole in Postmenopausal Women With Breast Cancer: Clinical Trial Safety and Pharmacodynamics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centro Nacional de Investigaciones Oncologicas CARLOS III (Other)
Collaborators: Dr. Miguel Angel Quintela Fandiño (CNIO) (Unknown); Dr, Ramón Colomer i Bosch (Unknown); FUNDACIÓN CRIS (Marta Cardona) as promotor (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNIO-BR-007
Record Dates: First submitted 2015-10-15; First posted 2015-12-02 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: breast cancer non metastatic; adjuvant letrozole; Nintedanib BIFF1120
MeSH Terms: conditions — Breast Neoplasms | interventions — nintedanib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Letrozole+Nintedanib (Experimental): Letrozole+Nintedanib
  Interventions: Drug: Nintedanib; Drug: Letrozole

INTERVENTIONS:
Drug: Nintedanib — Tablets of 100 mg. or 150 mg.
  Other Names: BIFF 1120
Drug: Letrozole — Tablet of 2.5 mg.

SUMMARY:
Open, multicenter phase I with gradual increase in dosage to evaluate the safety and tolerability of orally administered nintedanib plus letrozole orally (2.5 mg / day) for patients with breast cancer. Nintedanib is administered twice a day orally for 28 consecutive days (Days 1-28) in 4-week cycles.

DETAILED DESCRIPTION:
Phase 0 / I:

At level 1 it includes three patients. If any patient suffers dose limiting toxicity (DLT), it proceeds to the increase in dose to the next level. If 2/3 patients experience DLT, he will close the increased dose and extended / investigate the previous dose level with 3 additional patients.

If the level 2, but less than 1/3 the minimum of 6 patients experience TLD is reached, the phase I be suspended because not expected another rise above Level 2.

Dose levels:

* Level 1: Nintedanib 150 mg twice daily + oral letrozole 2.5 mg / day orally, in a cycle of 28 days.
* Level 2: Nintedanib 200 mg twice daily via oral + letrozole 2.5 mg / day orally, in a cycle of 28 days.
* At least the first cycle will be administered during Phase I. A total of six four-week cycles were administered at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Form signed informed consent.
2. Women ≥ 18 years.
3. Confirmed diagnosis of invasive non-metastatic breast cancer positive for hormone receptors. The inclusion of patients with ductal or lobular histology allowed.
4. Size greater than 1 cm tumor and any N or N ≥ 1 and any T, including inflammatory breast cancer.
5. Absence of metastatic involvement.
6. Postmenopausal state. Postmenopausal status is defined as more than 24 months after the last menstrual period, or previous known ovariectomy, or chemical, determined by FSH, LH and estradiol 17-B according to the local laboratory values over 12 months without menstruation.
7. ECOG performance status of 0 or 1
8. At least one month after the end of radiotherapy and / or chemotherapy.
9. At least 6 weeks since major surgery.
10. Patients currently treated with letrozole less than 6 months.
11. Primary surgery for breast cancer already done. The elderly women with advanced local or regional tumors in which hormone treatment is administered as monotherapy, regardless of the intent of the surgery are not candidates.
12. LVEF> 50%
13. Renal function, liver and adequate hematologic, defined by the following analytical results within 14 days prior to randomization or registration:

    * Absolute granulocyte count> 1.5 x 109 / L
    * Absolute platelet count> 100 x 109 / L
    * Hemoglobin> 10 g / dl
    * Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance> 50 ml / min
    * Serum bilirubin <1.25 ULN
    * AST / ALT ≤ 1.5 times the LS
14. Toxicities associated with chemotherapy recovery lesser extent 2 not tolerable.
15. Life expectancy> 6 months.

Exclusion Criteria:

1. HER2 overexpression defined as positive by immunohistochemistry HER-2-positive 2+ 3+ or FISH / CISH.
2. Absence of tumor tissue file.
3. T1 N0 stage patients are excluded.
4. Malignancy concomitant active, or diagnosis of another malignancy within the last five years, apart from non-melanoma or ductal / tubular breast carcinoma skin cancer (not received hormone treatment) or in situ cervical cancer, carcinoma colon in situ treated properly, as well as any diagnosis of tumor less than five years before the inclusion unsigned progression today.
5. Women of childbearing potential.
6. Pretreatment nintedanib. Use of other investigational drugs during the administration of adjuvant or neoadjuvant treatment is not an exclusion criterion as long as toxicity recovers.
7. Medical Condition concomitant serious, like eg myocardial infarction within 6 uncontrolled prior to inclusion in the study months, congestive heart failure, unstable angina, cardiomyopathy active, unstable ventricular arrhythmia, hypertension (according to the criteria of the NYHA) , psychotic disorders uncontrolled severe active infections, active peptic ulcer disease, psychiatric disease, HIV infection, active hepatitis, COPD or any other medical condition that might be aggravated by treatment or limits compliance.
8. Inability to make oral, or history of malabsorption syndrome medication.
9. Failure to comply with the study and follow-up procedures.
10. Anticoagulant therapy (except low-dose heparin or heparin washing as needed to maintain a permanent intravenous device) or antiplatelet therapy (except low-dose therapy with aspirin, less than 325 mg daily).
11. History of thromboembolic or hemorrhagic episodes that are clinically relevant in the past 6 months or hereditary predisposition to bleeding or thrombosis.
12. Contraindication to hormonal blockade or absence of hormone-blocking prescription from your doctor for any reason. Metastatic breast cancer or non-surgical (including inflammatory).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | 1-6 months
  Classified according to the version 4.03 of CTCAE criteria NCI1

SECONDARY OUTCOMES:
Evaluating FGFR1 modulation and inhibition levels of 17-B Estradiol | 1-6 months
  Assess the pharmacodynamic modulation of FGFR1 and inhibition levels of 17-B: determine plasma levels of FGF 23 ang 17- B estradiol (pg/mL)
Pharmacokinetic interactions | 29 days
  Determine the pharmacokinetic interactions nintedanib combined with letrozole: determine plasma levels of Nintedanib and Letrozole at day 0, day 15 and day 29 (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Cardona, Study Chair — Fundacion CRIS de Investigación para Vencer el Cáncer
Locations (3):
- Spain (3):
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital de La Princesa, Madrid
  - Clínica Quirón, Madrid

REFERENCES:
- [Derived] Quintela-Fandino M, Apala JV, Malon D, Mouron S, Hornedo J, Gonzalez-Cortijo L, Colomer R, Guerra J. Nintedanib plus letrozole in early breast cancer: a phase 0/I pharmacodynamic, pharmacokinetic, and safety clinical trial of combined FGFR1 and aromatase inhibition. Breast Cancer Res. 2019 May 24;21(1):69. doi: 10.1186/s13058-019-1152-x. PMID 31126332